CLINICAL TRIAL: NCT04027140
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the M/L Taper With Kinectiv Technology Stems and Necks
Brief Title: MDR - M/L Taper With Kinectiv Technology Stems and Necks
Status: Terminated | Type: Observational
Why Stopped: Zimmer Biomet no longer intends to market the M/L Taper with Kinectiv in the European Union and therefore has terminated study MDRG2017-89MS-56H.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-56H
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Hip Disease; Hip Fractures; Hip Injuries; Hip Arthritis; Hip Pain Chronic
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: M/L Taper with Kinectiv Technology Stems and Necks — Patients that have been implanted with a M/L Taper with Kinectiv Technology Stem and/or neck to repair hip malfunction/disease.

SUMMARY:
The objective of this consecutive series PMCF study is to collect data confirming safety, performance and clinical benefits of the M/L Taper with Kinectiv Technology Stems and Necks when used for primary or revision total hip arthroplasty (implants) at 1,2,5 and 10-year follow-up*. ML Taper with Kinectiv Technology has been on the market since 2008, but has insufficient long term clinical data. Therefore, a prospective aspect to the study will be necessary to reach the 10-year time point.

DETAILED DESCRIPTION:
The objective of this consecutive series PMCF study is to collect data confirming safety, performance and clinical benefits of the M/L Taper with Kinectiv Technology Stems and Necks when used for primary or revision total hip arthroplasty (implants) at 1,2,5 and 10-year follow-up*. ML Taper with Kinectiv Technology has been on the market since 2008, but has insufficient long term clinical data. Therefore, a prospective aspect to the study will be necessary to reach the 10-year time point.

The primary objective is to confirm safety of the study products. This will be assessed by recording the incidence and frequency of revisions, complications, and adverse events. Relationship of the events to either implant or instrumentation should be specified.

The secondary objective is the assessment of performance and clinical benefits by analyzing recorded patient-reported clinical outcomes measures (PROMs).

*Follow-up with the patient at the 10 year time point will be collected by the site prospectively and the 1, 2 and 5 year time point data will be collected by the sponsor retrospectively from an existing database including ML Taper with Kinectiv Technology patients from a Zimmer Biomet hip registry.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older
* Rheumatoid arthritis
* Osteoarthritis
* Traumatic arthritis
* Polyarthritis
* Collagen disorders
* Avascular necrosis of the femoral head
* Nonunion of previous fractures of the femur
* Acute femoral neck fractures
* Congenital hip dysplasia
* Protrusio acetabuli
* Previously failed endoprostheses
* Patient must be willing and able to sign IRB/EC approved informed consent.

Exclusion Criteria:

* Skeletal immaturity
* Loss of abductor musculature in the affected limb
* Poor bone stock (e.g., steroid-induced metabolic bone disease)
* Poor skin coverage around the hip joint
* Neuromuscular disease (e.g., Charcot's joint) in the affected limb
* Local and/or overt systemic infection
* Patient with a stove-pipe femur
* Stem implanted using cement fixation.
* Off-label use
* Uncooperative patient or patient with neurologic disorders who are incapable of following directions
* Patient is known to be pregnant or nursing
* Patient is a prisoner
* Patient is a known alcohol or drug abuser
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent Patient is unwilling to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of subjects implanted with a M/L Taper with Kinectiv Technology Stem and or Neck according to the approved indications
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-11-05 (Actual)

PRIMARY OUTCOMES:
Device safety assessed through the frequency and incidence of revisions, complications and adverse events | Out to 10 Years.
  The primary objective of this study is the assessment of the safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications, and adverse events. Relation of the events to either implant or instrumentation should be specified.
Device safety assessed through radiographic assessments | Out to 10 Years
  The primary objective of this study is to assess the safety of the device by reviewing radiographic data post implantation for each patient. A radiograph will be taken at each follow-up time point and reviewed by the surgeon to assess the frequency and incidence of any device related issues that may show up.

SECONDARY OUTCOMES:
Device Performance and Benefits evaluated through the Harris Hip Score outcome measure. | Out to 10 Years
  The HHS is divided into 4 sub-categories; pain (44 points), function (47 points), range of motion (5 points), and absence of deformity (4 points). Patients select a discrete set of answers which correspond to predefined point allocations based on the category. To obtain a final score, these values are summed.
Device Performance and Benefits evaluated through the EuroQolo Five Dimensions Questionnaire (EQ5D) outcome measure. | Out to 10 Years
  The EQ-5D measures 5 dimensions of general health; mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with a total of 5 questions. It is accompanied by the patient's self-assessment with the VAS. There are three versions of the EQ-5D; 3 level (3L), 5 level (5L), and a youth (Y) version based off of the 3L model.
  Each dimension is assigned one of three discrete levels for evaluation on the day of administration for the three level evaluation:
  Level 1 - No problems, no disability Level 2 - Some problems, moderate disability Level 3 - A lot of problems, severe disability
  The final score is a five digit composite of the responses ranging between 33333 - 11111 with 243 possible combinations in between for the 3L test. The 5L test can measure 3,125 different health states and ranges between 55555-11111.

CONTACTS AND LOCATIONS:
Overall Officials: Lynsey Boyle, Study Director — Zimmer Biomet
Locations (1):
- Orthopedic and Fracture Specialists, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No